CLINICAL TRIAL: NCT03350334
Title: Perioperative Duloxetine for Pain Management After Laparoscopic Hysterectomy: A Prospective Randomized Placebo-controlled Study
Brief Title: Perioperative Duloxetine for Pain Management After Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Ozguc Takmaz, M.D.,Assist. Prof, Department of Obstetrics and Gynecology, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ob&Gyn Maslak
Record Dates: First submitted 2017-11-13; First posted 2017-11-22 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Laparoscopic Hysterectomy; Postoperative Recovery; Postoperative Pain
Keywords: Duloxetine; laparoscopic hysterectomy; postoperative pain; postoperative recovery
MeSH Terms: conditions — Pain, Postoperative | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Prospective randomised
Who Masked: Participant
Masking Description: Participants do not know whether they take placebo or Duloxetine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Duloxetine (Active Comparator): The patients who will be given 60 mg duloxetine 2 hours before surgery and 24 hours after surgery.
  Interventions: Drug: Duloxetine
- Placebo Control (Placebo Comparator): The patients who will be given 60 mg placebo 2 hours before surgery and 24 hours after surgery.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Duloxetine — Peri-operative Duloxetine administration
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: placebo — Placebo administration
  Arms: Placebo Control

SUMMARY:
The aim of the investigators of the study is to evaluate the effect of peri-operative duloxetine on post-operative recovery in patients undergoing laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Patients with benign gynecologic conditions (fibroids, pelvic pain, uterine prolapse) who are planned to undergo laparoscopic hysterectomy will be enrolled in the study. After randomization, the study participants will be given 60 mg duloxetine 2 hours before surgery and 24 hours after surgery, whereas the control participants will be given placebo tablets.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign gynecologic conditions (fibroids, pelvic pain, uterine prolapse) who are planned to undergo laparoscopic hysterectomy will be enrolled in the study

Exclusion Criteria:

* Patients with chronic non-gynecologic conditions (liver or pulmonary disease, diabetes), using psychiatric drugs (anti-depressants, neuroleptics, lithium) in the last 1 year, those with duloxetine allergy, and patients using opioids for gynecologic or non-gynecologic conditions will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-03-10 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery-40 questionnaire total score | 24 hours after surgery
  Total scores of the Quality of Recovery-40 scale will be obtained 24 hours after surgery. Quality of Recovery-40 scale is a validated post-operative recovery questionnaire that consists of 40 questions, and 5 sub-components for pain (7), physical comfort (12), physical independence (5), emotional state (9), and psychological support (7). Positive items are scored from 1 (worst) to 5 (best); scores are reversed for negative items. Each item is scored ranging from 1 to 5. Total questionnaire score is calculated by sum of all items, and also sub-components by the sum of corresponding items. The total score ranges from 40 to 200.

SECONDARY OUTCOMES:
Narcotic analgesic consumption doses | 24 hours after surgery
  Number of total narcotic analgesic consumption doses of the participants through the post-operative 24 hours.
Length of hospital stay | post-operative 1 week
  number of days participants stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mete Gungor, MD,Prof, Study Chair — Acibadem Maslak Hospital
Locations (1):
- Acibadem Maslak Hospital, Sarıyer, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD sharing plan will be made at the end of the study

REFERENCES:
- [Result] Castro-Alves LJ, Oliveira de Medeiros AC, Neves SP, Carneiro de Albuquerque CL, Modolo NS, De Azevedo VL, De Oliveira GS Jr. Perioperative Duloxetine to Improve Postoperative Recovery After Abdominal Hysterectomy: A Prospective, Randomized, Double-Blinded, Placebo-Controlled Study. Anesth Analg. 2016 Jan;122(1):98-104. doi: 10.1213/ANE.0000000000000971. PMID 26421810
- [Result] YaDeau JT, Brummett CM, Mayman DJ, Lin Y, Goytizolo EA, Padgett DE, Alexiades MM, Kahn RL, Jules-Elysee KM, Fields KG, Goon AK, Gadulov Y, Westrich G. Duloxetine and Subacute Pain after Knee Arthroplasty when Added to a Multimodal Analgesic Regimen: A Randomized, Placebo-controlled, Triple-blinded Trial. Anesthesiology. 2016 Sep;125(3):561-72. doi: 10.1097/ALN.0000000000001228. PMID 27387351
- [Result] Ho KY, Tay W, Yeo MC, Liu H, Yeo SJ, Chia SL, Lo NN. Duloxetine reduces morphine requirements after knee replacement surgery. Br J Anaesth. 2010 Sep;105(3):371-6. doi: 10.1093/bja/aeq158. Epub 2010 Jun 23. PMID 20573635
- [Result] Wong K, Phelan R, Kalso E, Galvin I, Goldstein D, Raja S, Gilron I. Antidepressant drugs for prevention of acute and chronic postsurgical pain: early evidence and recommended future directions. Anesthesiology. 2014 Sep;121(3):591-608. doi: 10.1097/ALN.0000000000000307. PMID 25222675
- [Result] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540